CLINICAL TRIAL: NCT03757299
Title: Promoting Comprehensive Cervical Cancer Prevention and Better Women Health in Cameroon
Acronym: PCCCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Patrick Petignat (Other)
Responsible Party: Sponsor-Investigator, Prof. Patrick Petignat, Director of the gynecology departement, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017-01110
Record Dates: First submitted 2018-11-14; First posted 2018-11-28 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Human Papillomavirus DNA Tests; Papanicolaou Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self HPV (Experimental)
  Interventions: Diagnostic Test: HPV Test

INTERVENTIONS:
Diagnostic Test: HPV Test — Vaginal specimens for HPV test will be collected by participants themselves using flocked swabs after explanations by co-investigators. Two transport mediums will be used for those self-collected vaginal samples: NaCl 0.9%.
  Other Names: VIA/VILI,; Pap smear,; Cervical biopsy; ECC

SUMMARY:
In sub-Saharan Africa, cervical cancer is the leading cause of cancer death among women because of the difficulty in implementing screening programs. The main obstacles in these countries are poverty, lack of healthcare infrastructures and trained practitioners. With the availability of new technologies, researchers are looking for new strategies adapted to low- and middle-income countries to identify cervical precancerous lesions.

Current evidence shows that Human Papilloma Virus (HPV) testing is more effective than cytology (Pap smear) for cervical cancer screening in resource-limited settings. Indeed, the GeneXpert® HPV test offers the opportunity to prevent cervical cancer (CC) in a single visit: rapid detection of high-risk HPV (HPV) infection followed by same day treatment of HPV-positive women during the same visit (screen-and-treat approach).

However only a small proportion of HPV-positive women will develop cervical (pre)cancer, making it important to select those to treat. This triage can be achieved by colposcopy, cytology and visual inspection after application of acetic acid (VIA). Though VIA is the triage test recommended by WHO for resource-limited countries, it has not yet been widely assessed in sub-Saharan Africa (SSA).

The main objective of the investigators is to assess the performance of HPV-test followed by Visual Inspection after application of Acetic acid and Lugol's iodine VIA/VILI to detect cervical precancerous lesions in a screen-and-treat strategy in Cameroon (sub-Saharan Africa) where there is no cervical cancer-screening program.

The investigators organized a successful free screening campaign in Cameroon in 2015 that allowed to identify the expectations of women and their eagerness to benefit from prevention of gynecological cancers and sexually transmitted diseases.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 30-49 years, able to comply with the study protocol

Exclusion Criteria:

* Pregnancy
* Previous total hysterectomy
* Conditions impairing examination of the cervix

Ages: 30 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only women will be recruited by the study
Enrollment: 4473 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2024-07-09 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of HPV test followed by VIA/VILI to detect cervical precancerous lesions in sub-Saharan Africa using histology as gold standard | 3 - 5 years
  VIA/VILI is assessed by pelvic examination and Sensitivity and specificity are measured by using histology as gold stantard

SECONDARY OUTCOMES:
Prevalence of HPV infection | 3 - 5 years
  HPV self-test analysed by GeneXpert machine
Prevalence of cervical pre-cancer and cancer among Cameroonian women | 3 - 5 years
  Histological analyses of cervical biopsies and endocervical brushing
HPV clearance | 3 - 5 years
  Measured by self HPV performed at 6 and 12 months follow up
Persistance of CIN2+ disease at the 12-month follow-up | 3 - 5 years
  Histological analyses of cervical biopsies and endocervical brushing
Provide teaching material for professional training on cervical cancer prevention through VIA/VILI (cervical images database) | 3 - 5 years
  images database
Acceptability rate of self-HPV test and cervical cancer screening procedures | 3 years
  To assess the acceptability of self-HPV, patients complete a questionnaire comprising different questions about the collection device (embarassment, comfort, anxiety and confidence about the test).
  Likert Scale 4 points : 1 (not at all) to 4 (very).
Proportion of side effects and complications after thermoablation or LEEP | 3 - 5 years
  questionnaire
VIA test-positive rate (HPV-positive women); | 3 - 5 years
  VIA/VILI is assessed by pelvic examination
VIA test-positive rate after 1- year follow-up of VIA-negative tests | 3 - 5 years
  VIA/VILI is assessed by pelvic examination
Thermal ablation efficacy rate | 3 - 5 years
  Thermal ablation efficacy rate will be assessed according to the biopsy proven CIN2+ rate after thermoablation treatment at the 6 and 12-month follow-up. The absence of CIN2+ will determine the success of the treatment in a patient who previously had a CIN2+ lesion.
  Adverses event : bleeding, complications, hospitalization
Acceptability rate of thermoablation | 3 years
  To assess the acceptability of thermoablation, patients completed a questionnaire comprising different questions about treatment tolerance, pain and following side effects. Respondent were invited to rate answers on a likert scale of 1 (no accpetability) to 4 (high acceptability)
Sexual dysfunction score, score of anxiety and method of contraception after screening procedures, | 2 years
  SF12, Asex, STAI 6 Y-form
Number of women screened with and without community health care workers. | 2 years
  community health workers registre
Increase awareness on gynecological pathologies, including cervical cancer, sexually transmitted diseases and HIV, vaginal fistula in the community of the study area, | 3-5 years
  questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- University of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sormani J, Moukam A, Wisniak A, Yakam V, Schmidt NC, Kenfack B, Petignat P. Psychological and sexual impact of human papillomavirus screening in women in Cameroon: a prospective cohort study. BMC Womens Health. 2025 Dec 19;25(1):602. doi: 10.1186/s12905-025-04083-6. PMID 41420163
- [Derived] Broquet C, Vassilakos P, Ndam Nsangou FM, Kenfack B, Noubom M, Tincho E, Jeannot E, Wisniak A, Petignat P. Utility of extended HPV genotyping for the triage of self-sampled HPV-positive women in a screen-and-treat strategy for cervical cancer prevention in Cameroon: a prospective study of diagnostic accuracy. BMJ Open. 2022 Dec 22;12(12):e057234. doi: 10.1136/bmjopen-2021-057234. PMID 36549727
- [Derived] Petignat P, Kenfack B, Wisniak A, Saiji E, Tille JC, Tsuala Fouogue J, Catarino R, Tincho E, Vassilakos P. ABCD criteria to improve visual inspection with acetic acid (VIA) triage in HPV-positive women: a prospective study of diagnostic accuracy. BMJ Open. 2022 Apr 4;12(4):e052504. doi: 10.1136/bmjopen-2021-052504. PMID 35379615
- [Derived] Metaxas T, Kenfack B, Sormani J, Tincho E, Lemoupa Makajio S, Wisniak A, Vassilakos P, Petignat P. Acceptability and safety of thermal ablation to prevent cervical cancer in sub-Saharan Africa. BMC Cancer. 2022 Feb 2;22(1):132. doi: 10.1186/s12885-022-09202-2. PMID 35109806